CLINICAL TRIAL: NCT04398160
Title: Influence of Bilateral Cervical Manipulation (C3/C4) on Thoracoabdominal Kinematics on Healthy Young Adults: Randomized Controlled Trial (RCT)
Brief Title: Bilateral Cervical Manipulation (C3/C4) on Thoracoabdominal Kinematics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, Professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OST1-003
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Cervical manipulation; Osteopathic manual therapy; Thoracoabdominal kinematics; Qualisys system

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HVLA manipulation (Experimental): In the intervention of the experimental group, the investigator will be primarily on the right side of the volunteer and identify C3 through the cervical reference of jaw angle, which is at the disc level between C2/C3 and then contact with the phalanges of third metacarpal in the left transverse of this vertebra.
  The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally.
  Interventions: Other: HVLA C3/C4 manipulation
- Sham technique (Sham Comparator): The investigator will be primarily on the right side of the volunteer and identify the C3 vertebra, having as anatomical reference the angle of the jaw, which is at the disc level between C2/C3 and then contact, with the phalanges of the third metacarpal, the left transverse apophysis of this vertebra.
  The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally.
  Interventions: Other: Sham technique
- No intervention group (No Intervention): The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally.

INTERVENTIONS:
Other: HVLA C3/C4 manipulation — The investigator will apply an anterior and lateral translation associated with extension, homolateral inclination and contralateral rotation of the cervical. This procedure will increase the tension of the soft tissues to reduce the remaining slack and, finally, the thrust will be applied in pure rotation. Subsequently the head of the volunteer will be repositioned in the neutral position without applying any pressure and will wait 10 seconds in this position. Finally, the previous procedure will be repeated to the opposite side.
  Arms: HVLA manipulation
Other: Sham technique — The investigator will apply an anterior and lateral translation associated with extension, homolateral inclination and contralateral rotation of the cervical until the perception of tissue tension at the point of contact, holding this position for 10 seconds. The investigator then repositions the head of the volunteer in the neutral position without applying pressure, holding again this position for 10 seconds. Finally, the previous procedure will be repeated for the opposite side.
  Arms: Sham technique

SUMMARY:
There is evidence of the interdependence between the diaphragm and the C4 vertebral level with regard to nerve, fascial and muscular connections. The purpose of this study is to evaluate the influence of cervical bilateral manipulation (C3/C4) on the thoracoabdominal kinematics in healthy young adults.

DETAILED DESCRIPTION:
Due to respiration the thoracoabdominal kinematics is considered a complex mechanism that evolves the movement of the ribs and fascia, the diaphragmatic function, the respiratory muscles and the mechanical properties of the airways that includes a coordinated reflex neural activity. The phrenic nerve (C3 to C5) is responsable for the motor and sensory innervation of the diaphragm.

The High Velocity Low Amplitude (HVLA) vertebral manipulation stimulates the corresponding spinal nerves. It is well known that when this manipulation is applied to cervical region induces vasomotor cutaneous and cardiorespiratory modifications in autonomic nervous system.

The sample composed of healthy young adults (aged 18-40 years) will be assigned randomly in three groups: experimental group (bilateral C3/C4 HVLA manipulation), sham manipulation group (passive cervical mobilization) and control group (no intervention). The thoracoabdominal kinematics measures will be assessed at baseline, right after the intervention and five minutes after the second measure using the Qualisys Motion Capture System.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 18 and 40 years of age.

Exclusion Criteria:

* Attending a degree in Osteopathy or being a health professional in this area;
* Apprehension to cervical manipulation;
* Be pregnant;
* Presenting cervical pain on the day of the study;
* Does not comply with the Australian Vertebral Artery Protocol guidelines;
* Having a clinical history of cervical and/or thoracoabdominal surgery;
* Having a clinical history of cervical trauma during the prior 12 months;
* Recurrent use of anti-coagulant and/or analgesic, muscle relaxant or anti-inflammatory therapeutics during the week before the study;
* Have been submitted to any manual intervention at cervical region during the week before the study;
* Having cardio-respiratory, neurological, rheumatic, oncologic and/or systemic diagnosed pathologies.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in anterior-to-posterior of the abdomen right after the intervention | Immediately after the intervention
  The Qualysis Motion Capture System will measure the variation of the tridimensional movement of the abdomen through the positioning of two reflectors that will be placed in standardized points: in the umbilicus and the spinal process of L3. The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally for 90 seconds.
  This measure instrument have eight infrared cameras which after the calibration process will determine the data of the tridimensional thoracoabdominal amplitude variations of the volunteer by the kinematic of the reflex markers.
Change from Baseline in anterior-to-posterior of the abdomen 5 minutes after the intervention | 5 minutes after the intervention
  The Qualysis Motion Capture System will measure the variation of the tridimensional movement of the abdomen through the positioning of two reflectors that will be placed in standardized points: in the umbilicus and the spinal process of L3. The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally for 90 seconds.
  This measure instrument have eight infrared cameras which after the calibration process will determine the data of the tridimensional thoracoabdominal amplitude variations of the volunteer by the kinematic of the reflex markers.

SECONDARY OUTCOMES:
Change from Baseline in anterior-to-posterior of the upper ribcage right after the intervention | Immediately after the intervention
  The Qualysis Motion Capture System will measure the variation of the tridimensional movement of the abdomen through the positioning of two reflectors that will be placed in standardized points: in the xiphoid process of sternum and the spinal process of seventh thoracic vertebra (T7). The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally for 90 seconds).
  This measure instrument have eight infrared cameras which after the calibration process will determine the data of the tridimensional thoracoabdominal amplitude variations of the volunteer by the kinematic of the reflex markers.
Change from Baseline in medial-to-lateral of the lower ribcage right after the intervention | Immediately after the intervention
  The Qualysis Motion Capture System will measure the variation of the tridimensional movement of the abdomen through the positioning of two reflectors that will be placed in standardized points: in the alignment of the mid-axillar line with the ninth rib bilaterally. The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally for 90 seconds.
  This measure instrument have eight infrared cameras which after the calibration process will determine the data of the tridimensional thoracoabdominal amplitude variations of the volunteer by the kinematic of the reflex markers.
Change from Baseline in anterior-to-posterior of the upper ribcage 5 minutes after the intervention | 5 minutes after the intervention
  The Qualysis Motion Capture System will measure the variation of the tridimensional movement of the abdomen through the positioning of two reflectors that will be placed in standardized points: in the xiphoid process of sternum and the spinal process of seventh thoracic vertebra (T7). The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally for 90 seconds.
  This measure instrument have eight infrared cameras which after the calibration process will determine the data of the tridimensional thoracoabdominal amplitude variations of the volunteer by the kinematic of the reflex markers.
Change from Baseline in medial-to-lateral of the lower ribcage 5 minutes after the intervention | 5 minutes after the intervention
  The Qualysis Motion Capture System will measure the variation of the tridimensional movement of the abdomen through the positioning of two reflectors that will be placed in standardized points: in the alignment of the mid-axillar line with the ninth rib bilaterally. The volunteer will be seated with 110º of hip and knee flexion using a digital goniometer and will be asked to breath normally for 90 seconds.
  This measure instrument have eight infrared cameras which after the calibration process will determine the data of the tridimensional thoracoabdominal amplitude variations of the volunteer by the kinematic of the reflex markers.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Tecnologia da Saúde do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Siribumrungwong K, Sinchai C, Tangtrakulwanich B, Chaiyamongkol W. Reliability and Accuracy of Palpable Anterior Neck Landmarks for the Identification of Cervical Spinal Levels. Asian Spine J. 2018 Feb;12(1):80-84. doi: 10.4184/asj.2018.12.1.80. Epub 2018 Feb 7. PMID 29503686
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] Hutting N, Kerry R, Coppieters MW, Scholten-Peeters GGM. Considerations to improve the safety of cervical spine manual therapy. Musculoskelet Sci Pract. 2018 Feb;33:41-45. doi: 10.1016/j.msksp.2017.11.003. Epub 2017 Nov 3. PMID 29153924
- [Background] Kranenburg HA, Schmitt MA, Puentedura EJ, Luijckx GJ, van der Schans CP. Adverse events associated with the use of cervical spine manipulation or mobilization and patient characteristics: A systematic review. Musculoskelet Sci Pract. 2017 Apr;28:32-38. doi: 10.1016/j.msksp.2017.01.008. Epub 2017 Jan 23. PMID 28171776
- [Background] de Camargo VM, Alburquerque-Sendin F, Berzin F, Stefanelli VC, de Souza DP, Fernandez-de-las-Penas C. Immediate effects on electromyographic activity and pressure pain thresholds after a cervical manipulation in mechanical neck pain: a randomized controlled trial. J Manipulative Physiol Ther. 2011 May;34(4):211-20. doi: 10.1016/j.jmpt.2011.02.002. Epub 2011 Mar 21. PMID 21621722
- [Background] Moser N, Mior S, Noseworthy M, Cote P, Wells G, Behr M, Triano J. Effect of cervical manipulation on vertebral artery and cerebral haemodynamics in patients with chronic neck pain: a crossover randomised controlled trial. BMJ Open. 2019 May 28;9(5):e025219. doi: 10.1136/bmjopen-2018-025219. PMID 31142519
- [Background] Bordoni B, Marelli F. The fascial system and exercise intolerance in patients with chronic heart failure: hypothesis of osteopathic treatment. J Multidiscip Healthc. 2015 Oct 30;8:489-94. doi: 10.2147/JMDH.S94702. eCollection 2015. PMID 26586951
- [Result] Goyal M, Goyal K, Narkeesh K, Samuel AJ, Arumugam N, Chatterjee S, Sharma S. Efficacy of Osteopathic Manipulative Treatment Approach in the Patient with Pulmonary Fibrosis in Critical Care Outpatient Department. Indian J Crit Care Med. 2017 Jul;21(7):469-472. doi: 10.4103/0972-5229.210648. PMID 28808371
- [Result] Taylor HH, Murphy B. Altered sensorimotor integration with cervical spine manipulation. J Manipulative Physiol Ther. 2008 Feb;31(2):115-26. doi: 10.1016/j.jmpt.2007.12.011. PMID 18328937
- [Result] Perry J, Green A, Singh S, Watson P. A preliminary investigation into the magnitude of effect of lumbar extension exercises and a segmental rotatory manipulation on sympathetic nervous system activity. Man Ther. 2011 Apr;16(2):190-5. doi: 10.1016/j.math.2010.10.008. Epub 2010 Nov 23. PMID 21106433
- [Result] Mesquita Montes A, Tam C, Crasto C, Argel de Melo C, Carvalho P, Santos R, Vilarinho R, Vilas-Boas JP. Forward trunk lean with arm support affects the activity of accessory respiratory muscles and thoracoabdominal movement in healthy individuals. Hum Mov Sci. 2018 Oct;61:167-176. doi: 10.1016/j.humov.2018.07.011. Epub 2018 Aug 11. PMID 30107366
- [Result] Anderst WJ, Gale T, LeVasseur C, Raj S, Gongaware K, Schneider M. Intervertebral kinematics of the cervical spine before, during, and after high-velocity low-amplitude manipulation. Spine J. 2018 Dec;18(12):2333-2342. doi: 10.1016/j.spinee.2018.07.026. Epub 2018 Aug 22. PMID 30142458
- [Result] de Camargo VM, Alburquerque-Sendín F, Bérzin F, Stefanelli VC, Rodrigues Pedroni C, & Santos K. Immediate Effects of the Ashmore Manipulation Technique C5/C6, in Muscle Activity in patients with Mechanical Neck Pain. European Journal Osteopathy & Clinical Related Research, 2012; 7(1), 2-9.